CLINICAL TRIAL: NCT01250886
Title: Intravenous Fluid Administration in Patients Undergoing Colonoscopy: Double Blind, Randomised Clinical Trial of Underlying Acid-base Derangement
Brief Title: Acid-base Balance in Patients Undergoing Colonoscopy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Phongthara Vichitvejpaisal", Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 456/2553(EC2)
Record Dates: First submitted 2010-11-29; First posted 2010-12-01 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Colonoscopy; Bowel Preparation
MeSH Terms: interventions — Ringer's Lactate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Normal saline solution (Placebo Comparator): Blood sample is obtained from patient in either forearm immediately before a Normal saline solution administered on the same site. The volume of fluid administration is calculated by means of Holliday and Segar formula.
  Interventions: Drug: Normal saline solution
- Lactated Ringer's solution (Active Comparator): Lactated Ringer's solution is administered. The volume of fluid administration is calculated by means of Holliday and Segar formula.
  Interventions: Drug: Lactated Ringer's solution
- Acetate Ringer's solution (Active Comparator): Acetate Ringer's solution is administered. The volume of fluid administration is calculated by means of Holliday and Segar formula.
  Interventions: Drug: Acetate Ringer's solution

INTERVENTIONS:
Drug: Lactated Ringer's solution — Lactated Ringer's solution is administered. The volume of fluid administration is calculated by means of Holliday and Segar formula.
  Other Names: LRS
  Arms: Lactated Ringer's solution
Drug: Normal saline solution — Normal saline solution is administered. The volume of fluid administration is calculated by means of Holliday and Segar formula.
  Other Names: NSS
  Arms: Normal saline solution
Drug: Acetate Ringer's solution — Acetate Ringer's solution is administered. The volume of fluid administration is calculated by means of Holliday and Segar formula.
  Other Names: ARS
  Arms: Acetate Ringer's solution

SUMMARY:
The purpose of this study is to determine whether fluid administration in patients undergoing colonoscopy should affect acid-base disorder in term of the strong ion differences.

DETAILED DESCRIPTION:
This is a prospective, double-blinded, randomized control trial. The study enrolls 90 consecutive outpatients, well-prepared bowel, scheduled to undergo routine colonoscopy for screening, surveillance, or diagnosis of colorectal diseases. At the outpatient clinic, the co-researcher invites patients who meet the inclusion criteria to join the study. The process of the project is explained to the interested patients in details before an informed consent is obtained and the first blood sample is conducted.

On the day of colonoscopy, all participants are randomized equally into three groups: Normal saline solution (NSS, n = 30) as control group, lactated Ringer's solution (LRS, n = 30) and acetated Ringer's solution (ARS, n = 30) as treatment groups. The second blood sample is obtained from patients via 20-gauge needle in either forearm immediately before an allocated intravenous (IV) fluid administered on the same site. The volume of fluid is calculated by means of Holliday and Segar formula.

The colonoscopy under total intravenous anesthesia is performed between 9:00 a.m. and 3:00 p.m. At the end of colonoscopy, the patients spontaneously wake up in the recovery room. After they gain conscious and all vital signs are stable; the intravenous fluid is off and the third blood sample is taken in the other forearm. After completion of the procedure, the patient is advised to follow the discharge instructions.

ELIGIBILITY:
Inclusion Criteria:

* male or non-pregnant
* non-lactating female out-patient scheduled for routine colonoscopy
* over 18 years of age
* eligible for taking PEG or NaP for bowel preparation, and willing to sign informed consent.

Exclusion Criteria:

* insulin-dependant diabetes
* renal insufficiency (creatinine >2.0 mg⁄ dL)
* renal dialysis
* uncontrolled congestive heart failure (American Heart Association Classification III or IV congestive heart failure)
* unstable angina
* untreated cardiac arrhythmia
* ileus and⁄or acute obstruction or perforation
* ileostomy
* presence of a colostomy
* history of a partial colon resection
* active gastrointestinal bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-12; Primary Completion 2015-10 (Actual); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Acid-base disorder as a Measure of Strong Ion Difference. | 3 days
  The strong ion difference (SID) is calculated by means of the differences between the positively and negatively charged strong ions in plasma. The strong ion difference affected by bowel preparation and intravenous fluid administration during colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Phongthara Vichitvejpaisal, M.D., Ph.D., Principal Investigator — Mahidol University